Fit Group Oneway Analysis of percent By Treatment



#### **Means and Std Deviations**

| Level | Number | Mean | Std Dev S | td Err Mean | Lower 95% | Upper 95% |
|---|---|---|---|---|---|---|
| Control | 11 | 24.136364 | 16.261935 | 4.903158 | 13.211447 | 35.061281 |
| Test | 11 | <mark>19.118182</mark> | 10.566061 | 3.1857871 | 12.019806 | 26.216558 |

#### t Test Test-Control

Assuming unequal

| Difference<br>Std Err Dif<br>Upper CL Dif | -5.018 t Ratio<br>5.847 DF<br>7.309 Prob > t | -0.85821<br>17.16612<br><mark>0.4026</mark> |
|---|---|---|
| Lower CL Dif | -17.346 Prob > t | 0.7987 |
| Confidence | 0.95 Prob < t | 0.2013 |



# Oneway Analysis of RW changes By Treatment



#### **Means and Std Deviations**

| Level | Number | Mean | Std Dev S | Std Err Mean | Lower 95% | Upper 95% |
|---|---|---|---|---|---|---|
| Control | 11 | -0.813 | 0.5934787 | 0.1789406 | -1.211704 | -0.414296 |
| Test | 11 | -1.227818 | 0.9734682 | 0.2935117 | -1.881803 | -0.573833 |

#### t Test Test-Control

Assuming unequal variances

| Difference | -0.4148 t Ratio | -1.20672 |
|--------------|-------------------|----------|
| Std Err Dif | 0.3438 DF | 16.5313 |
| Upper CL Dif | 0.3120 Prob > t | 0.2445 |
| Lower CL Dif | -1.1417 Prob > t | 0.8777 |
| Confidence | 0.95 Prob < t | 0.1223 |



### Oneway Analysis of RH changes By Treatment



#### **Means and Std Deviations**

| Level | Number | Mean | Std Dev | Std Err<br>Mean | Lower 95% | Upper 95% |
|---|---|---|---|---|---|---|
| Control | 11 | -1.35 | 0.7771744 | 0.2343269 | -1.872113 | -0.827887 |
| Test | 11 | -1 | 0.7375636 | 0.2223838 | -1.495502 | -0.504498 |

#### t Test Test-Control Assuming unequal variances

Difference -0.3500 t Ratio -1.083412 Std Err Dif DF 0.3231 19.94552 Upper CL Dif Prob > |t|1.0240 0.2915 Lower CL Dif Prob > t-0.3240 0.1458Confidence 0.8542  $Prob \le t$ 

0.95



# **Control Group BPW:**

### **Bivariate Fit of RW Control By BPW**



# Linear Fit

RW = 1.0799645 - 0.1553762\*BBW

### **Summary of Fit**

| RSquare | 0.072206 |
|----------------------------|----------|
| RSquare Adj | -0.03088 |
| Root Mean Square Error | 0.602573 |
| Mean of Response | 0.813 |
| Observations (or Sum Wgts) | 11 |

# **Analysis of Variance**

| Source | DF | Sum of Squares | Mean Square | F Ratio |
|----------|----|----------------|-------------|----------|
| Model | 1 | 0.2543228 | 0.254323 | 0.7004 |
| Error | 9 | 3.2678472 | 0.363094 | Prob > F |
| C. Total | 10 | 3.5221700 | | 0.4243 |

#### **Parameter Estimates**

| Term | Estimate | Std Error | t Ratio | Prob> t |
|-----------|-----------|-----------|---------|---------|
| Intercept | 1.0799645 | 0.367097 | 2.94 | 0.0164* |
| BBW | -0.155376 | 0.185653 | -0.84 | 0.4243 |

# **Bivariate Fit of RH Control By BBW**



Linear Fit

### **Summary of Fit**

| RSquare | 0.816877 |
|----------------------------|----------|
| RSquare Adj | 0.79653 |
| Root Mean Square Error | 0.350565 |
| Mean of Response | 1.35 |
| Observations (or Sum Wgts) | 11 |

### **Analysis of Variance**

| Source | DF | Sum of Squares | Mean Square | F Ratio |
|----------|----|----------------|-------------|----------|
| Model | 1 | 4.9339386 | 4.93394 | 40.1474 |
| Error | 9 | 1.1060614 | 0.12290 | Prob > F |
| C. Total | 10 | 6.0400000 | | 0.0001* |

#### **Parameter Estimates**

| Term | Estimate | Std Error | t Ratio | Prob> t |
|-----------|-----------|-----------|---------|---------|
| Intercept | 2.5258657 | 0.21357 | 11.83 | <.0001* |
| BBW | -0.684366 | 0.108009 | -6.34 | 0.0001* |

### **Test Group BPW:**

### **Bivariate Fit of RW Test By BPW**



— Linear Fit

#### Linear Fit

RW = 1.0197564 + 0.1368009\*BPW

### **Summary of Fit**

| RSquare | 0.021005 |
|----------------------------|----------|
| RSquare Adj | -0.08777 |
| Root Mean Square Error | 1.015291 |
| Mean of Response | 1.227818 |
| Observations (or Sum Wgts) | 11 |

# **Analysis of Variance**

| Source | DF | Sum of Squares | Mean Square | F Ratio |
|----------|----|----------------|-------------|----------|
| Model | 1 | 0.1990565 | 0.19906 | 0.1931 |
| Error | 9 | 9.2773471 | 1.03082 | Prob > F |
| C. Total | 10 | 9.4764036 | | 0.6707 |

### **Parameter Estimates**

| Term | Estimate | Std Error | t Ratio | Prob> t |
|-----------|-----------|-----------|---------|---------|
| Intercept | 1.0197564 | 0.563814 | 1.81 | 0.1040 |
| BBW T | 0.1368009 | 0.311309 | 0.44 | 0.6707 |

# **Bivariate Fit of RH Test By BPW**



Linear Fit

# **Summary of Fit**

| RSquare | 0.150948 |
|----------------------------|----------|
| RSquare Adj | 0.056609 |
| Root Mean Square Error | 0.675152 |
| Mean of Response | 1.027273 |
| Observations (or Sum Wgts) | 11 |

# **Analysis of Variance**

| Source | DF | Sum of Squares | Mean Square | F Ratio |
|----------|----|----------------|-------------|----------|
| Model | 1 | 0.7293518 | 0.729352 | 1.6001 |
| Error | 9 | 4.1024663 | 0.455830 | Prob > F |
| C. Total | 10 | 4.8318182 | | 0.2377 |

### **Parameter Estimates**

| Term | Estimate | Std Error | t Ratio | Prob> t |
|-----------|-----------|-----------|---------|---------|
| Intercept | 1.4255382 | 0.374927 | 3.80 | 0.0042* |
| BBW T | -0.26186 | 0.207015 | -1.26 | 0.2377 |